CLINICAL TRIAL: NCT00751582
Title: Effective Means to Address Moderately Malnourished Children Within BINP Communities
Brief Title: Effective Means to Address Moderately Malnourished Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: World Bank (Other)
Responsible Party: Principal Investigator, ICDDRB
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 98-018
Record Dates: First submitted 2008-05-17; First posted 2008-09-12 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2008-09

CONDITIONS: Malnutrition
Keywords: nutrition; education; supplementation
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements; Nutrition Assessment; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Food supplementation and nutrition education
  Interventions: Dietary Supplement: Food supplementation and nutrition education; Other: Control Group
- 1 (Experimental): Nutrition Education only
  Interventions: Behavioral: Nutrition education

INTERVENTIONS:
Dietary Supplement: Food supplementation and nutrition education — Food supplementation and nutrition education for three months
  Other Names: PUSHTI PACKET
  Arms: 2
Behavioral: Nutrition education — Nutrition education for children for three months
  Other Names: PUSHTI PACKET
  Arms: 1
Other: Control Group — No Nutrition Education
  Arms: 2

SUMMARY:
Supplementary feeding and intensive IEC at the community level will effectively reduce moderate PEM compared to the control children within 3 months .

Intensive nutrition education at the household level will reduce by at least one third of the prevalence of moderate malnutrition (40% of present level) within a short period of 3 months

DETAILED DESCRIPTION:
Bangladesh is one of the countries having highest proportions of malnourished children in the world. The Bangladesh Integrated nutrition Project (BINP) is a recent initiative of the Government of Bangladesh to reduce malnutrition of women and children under two years of age. The BINP includes a specific programme to address severely malnourished children at the community level, however there is no such programme directed toward moderately malnourished children. Moderately malnourished children form a large proportion of children in the community, and with success of the BINP, this proportion is growing, as severely malnourished children shift to the moderately malnourished category. To address this, operations research will be undertaken in a BINP thana named Shahrasti, in Chandpur District over a 6 month period. A total of 300 children in three groups from Community Nutrition Centres (CNC) will be studied. There will be groups in the study. In addition to usual component of the BINP, mothers of the first group of intervention will receive intensive nutrition education and motivation for child care, complementary food demonstration, and household food mobilization for child feeding weekly for first four weeks then reinforced every two weeks. The second intervention group will receive a packet of the usual BINP food supplement daily for 6 days a week for 3 months and nutrition education at the same intensity. The third group will be a control group and will receive only the usual programme inputs of BINP and their weight gain will be recorded. The CNP, women group and village nutrition committee will be involved. Focus group discussion will be held with mothers. Data on morbidity will be collected and necessary medical advise will be given equal to each group. Data collection, counseling on child caring practice, food demonstration and nutrition education using IEC will be organized and supervised by project staff. It is assumed that if the intervention is successful, and once the nutritional status improves, they are likely to maintain good health. The IEC on dietary practice will be communicated to the village members for preventive measures. Data will be analyzed for change in nutrition groups from moderate to mild malnutrition or normal nutrition and will be compared between the control and two intervention groups. It is expected that the results of the study will help to address to reduce moderate malnutrition existing in the large proportion of malnourished children. This will in turn reduce the risk of regressing to severe malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Less than 2 years moderately malnourished children

Exclusion Criteria:

* Nourished children

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 1998-07; Primary Completion 1998-11 (Actual); Study Completion 1998-11 (Actual)

PRIMARY OUTCOMES:
Weight and length to assess nutritional status of the children | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Swapan K Roy, PhD, FRCP, Principal Investigator — Senior Scientist, ICDDR,B
Locations (1):
- ICDDRB, Dhaka, Bangladesh